CLINICAL TRIAL: NCT01902199
Title: Studying a Novel Intervention, the Tobacco Retraining of Automatic Approach (TRAA), to Treat Individuals With Tobacco Dependence and Severe Concurrent Disorders
Brief Title: Tobacco Retraining of Automatic Approach to Treat Individuals With Tobacco Dependence and Severe Concurrent Disorders.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Provincial Health Services Authority British Columbia (Other)
Responsible Party: Principal Investigator, Christian Schutz, Dr. Christian Schutz, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H13-01422
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Tobacco Retraining of Automatic Approach; Placebo Task

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- TRAA (Active Comparator): participants will be given the active TRAA intervention where landscape images are linked with a push motion, and portrait images linked with a pull motion. Pictures will exclusively be related to smoking.
  Interventions: Behavioral: TRAA intervention
- Control (Placebo Comparator): participants will be given a mix of landscape and portrait pictures, equally divided into push or pull. the images will be a mix of smoking related pictures and non smoking pictures.
  Interventions: Behavioral: TRAA intervention

INTERVENTIONS:
Behavioral: TRAA intervention — The Tobacco Retraining of Automatic Approach The tobacco-RAA will be the intervention in changing approach tendencies towards tobacco. The task uses pictures of tobacco related objects (e.g, a cigarette) and pictures of non-tobacco related objects (e.g, a spoon). Patients will be presented with a joystick while pictures are presented on a computer screen. Patients will be presented with pictures, pulling pictures in a portrait format, while they push pictures in a landscape format. In the experimental condition pictures pushed will almost exclusively be smoking related pictures. In the control condition smoking pictures will be equally divided into push and pull conditions.

SUMMARY:
A randomized control trial evaluating a novel smoking cessation intervention in individuals at a an inpatient clinic for clients with addiction and concurrent disorders. The intervention is based on cognitive bias modification, where participants are explicitly or implicitly trained to make avoidance movements by pushing a joystick in response to pictures of smoking, and as a result altering their cognitive biases towards smoking and tobacco dependence.

Hypothesis: Participation in the experimental (tobacco-avoidance) condition will induce reduction of smoking, assessed as lower levels of carbon monoxide measured at baseline and 12 week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Proficiency to read and write english
* A minimum score of 5 or higher on the fagerström test for nicotine dependence, indicating a medium dependence
* Current smoking will be validated by Carbon monoxide breath monitor

Exclusion Criteria:

* Patients not yet stabilized enough to allow for regular participation in the intervention

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Carbon monoxide levels in breath | baseline, 12 weeks
  The breath carbon monoxide monitoring device will be used both before the intervention for a baseline measure and at the 12-week follow-up for comparison. These two measurements will be used to detect changes in smoking patterns that may have occurred during this interval. The method allows to objectify abstinence from smoking.

SECONDARY OUTCOMES:
Fagerström test for Nicotine dependence (FTND) | Baseline
  The FTND is a 6-item questionnaire scored to test level of nicotine dependence, and will be presented to patients prior to the intervention. Patients meeting a cut-off score of 5 or higher will be eligible to participate in the intervention portion of this study.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Schutz, MD, Principal Investigator — UBC/ VCH
Locations (1):
- Burnaby Centre for Mental Health and Addiction, Burnaby, British Columbia, Canada